CLINICAL TRIAL: NCT02512900
Title: A Phase 1, Open-label Study to Evaluate the Pharmacokinetics of MEDI9929 (AMG 157) in Adolescents With Mild to Moderate Asthma
Brief Title: A Study to Evaluate the Pharmacokinetics of MEDI9929 (AMG 157) in Adolescents With Mild to Moderate Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D5180C00002; 2014-005450-19 (EudraCT Number)
Record Dates: First submitted 2015-07-24; First posted 2015-07-31 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab; Injections, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MEDI9929, 140 mg, Cohort 1 (12 to 14 years) (Experimental): On Day 1, one MEDI9929 subcutaneous injection of 70 mg was given into the anterior aspect of one thigh immediately followed by the second injection of 70 mg into the anterior aspect of the contralateral thigh to make the required dose of 140 mg in participants with 12 to 14 years of age.
  Interventions: Drug: MEDI9929, 140 mg
- MEDI9929, 140 mg, Cohort 2 (15 to 17 years) (Experimental): On Day 1, one MEDI9929 subcutaneous injection of 70 mg was given into the anterior aspect of one thigh immediately followed by the second injection of 70 mg into the anterior aspect of the contralateral thigh to make the required dose of 140 mg in participants with 15 to 17 years of age.
  Interventions: Drug: MEDI9929, 140 mg

INTERVENTIONS:
Drug: MEDI9929, 140 mg — On Day 1, two MEDI9929 subcutaneous injection of 70 mg each were given into the anterior aspect of one thigh immediately followed by the second injection into the anterior aspect of the contralateral thigh to make the required dose of 140 mg in participants of 12 to 17 years of age.
  Other Names: Subcutaneous single-dose

SUMMARY:
To evaluate the PK profile of a single-dose of 140 mg subcutaneous (SC) administration of MEDI9929 (AMG 157) in adolescent subjects with mild to moderate asthma.

DETAILED DESCRIPTION:
The primary objective is to evaluate the PK profile of a single-dose of 140 mg subcutaneous (SC) administration of MEDI9929 (AMG 157) in adolescent subjects with mild to moderate asthma. The secondary objective is to evaluate the safety and tolerability of MEDI9929 and to evaluate the immunogenicity of MEDI9929 (AMG 157). The exploratory objective is to evaluate the effect of MEDI9929 (AMG 157) on pulmonary function

ELIGIBILITY:
Inclusion Criteria

* Age 12 to 17 years (inclusive) at both screening and Day 1.
* Physician diagnosed asthma for a minimum of 6 months prior to screening.
* Physician prescribed daily use of asthma controller medication
* Prebronchodilator FEV1 of ≥ 70% of predicted normal value at screening.
* A postbronchodilator increase in FEV1 ≥ 12% and ≥ 200 mL at screening.
* If on allergen immunotherapy, subjects must be on a stable maintenance dose and schedule ≥ 1 month prior to Visit 1.
* Weight ≥ 30 kg at both screening and Day 1.
* Body mass index for age at both screening and Day 1 that is between 5th and 95th percentile
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use highly effective contraception from screening
* Nonsterilized males who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception from screening

Exclusion Criteria:

* History of a deterioration in asthma that required a burst of systemic corticosteroids within 3 months of screening, up to and including Day 1.
* Clinical characteristics at either screening or Day 1 that are consistent with uncontrolled asthma as described in GINA guideline.
* History of hospitalization (overnight admission) for asthma during the 6 months prior to screening.
* History of intubation for the management of a deterioration in asthma.
* History of systemic corticosteroid use for the maintenance treatment of asthma within 3 months prior to screening.
* History of allergy or reaction to any component of the investigational product formulation or history of anaphylaxis following any biologic therapy.
* Any active medical condition other than asthma, that in the opinion of the investigator and/or medical monitor, may compromise the safety of the subject in the study or interfere with evaluation of the investigational product or reduce the subject's ability to participate in the study (subjects with atopic skin conditions and allergic rhinitis are permitted).
* Pregnant or breastfeeding females.
* Current tobacco smoking or cessation of smoking for ≤ 6months prior to screening.
* Any clinically relevant abnormal findings which in the opinion of the investigator or medical monitor, may compromise the safety of the subject in the study or interfere with evaluation of the investigational product or reduce the subject's ability to participate in the study.
* Evidence of active liver disease,
* Positive hepatitis B or hepatitis C virus
* A positive human immunodeficiency virus (HIV) test at screening or subject taking antiretroviral medications
* Major surgery within 8 weeks prior to Visit 1, or planned in-patient surgery or hospitalization during the study period.
* History of any known primary immunodeficiency disorder
* History of a clinically significant infection
* A helminth parasitic infection within 24 weeks of Visit 1 that has not been treated or has not responded to standard of care therapy.
* History of cancer.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2016-05-17 (Actual); Study Completion 2016-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rene van der Merwe, MBChB, MSc, FFPM, Study Director — MedImmune LLC
Locations (3):
- Poland (3):
  - Research Site, Kielce
  - Research Site, Lodz
  - Research Site, Wroclaw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescent participants (12 to 17 years, inclusive) with mild to moderate asthma were recruited in an open-label fashion to receive a single-dose of MEDI9929 (also known as tezepelumab or AMG 157) at two study centers in Poland from Sep 2015 to May 2016.
Pre-assignment Details: A total of 26 participants were screened, out of these, 21 subjects were randomized and completed the study at 2 investigative sites in Poland.
Groups:
- MEDI9929, 140 mg, (12 to 14 Years); MEDI9929, 140 mg, (15 to 17 Years): On Day 1, a single dose of MEDI9929 was administered subcutaneously to all participants.
Period: Overall Study
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years) | TOTAL
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.5 (0.8) | 15.9 (0.7) | 14.7 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Zero to Infinity (AUC [0-infinity])
Description: The pharmacokinetic (PK) parameter AUC (0 to infinity) was estimated based on the serum concentrations of MEDI9929. Serum concentrations of MEDI9929 were measured by enzyme-linked immunosorbent assay.
Time Frame: Predose on Day 1 and Day 2, 4, 7, 11, 15, 22, 29, 43, 57 and 85 post-dose.
Population: PK Population: All participants who received MEDI9929 and have a sufficient number of serum concentration measurements for computing PK parameters.
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Number analyzed (Participants) | 11 | 10
μg*day/mL | 1020 (355) | 881 (185)

2. Primary Outcome: Area Under the Concentration-Time Curve From Zero to Last Observation (AUC [0-t])
Description: The PK parameter AUC (0-t) was estimated based on the serum concentrations of MEDI9929. Serum concentrations of MEDI9929 were measured by enzyme-linked immunosorbent assay.
Time Frame: Predose on Day 1 and Day 2, 4, 7, 11, 15, 22, 29, 43, 57 and 85 post-dose.
Population: PK Population
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Number analyzed (Participants) | 11 | 10
μg*day/mL | 906 (284) | 780 (171)

3. Primary Outcome: Dose-normalized AUC (0-infinity) (AUC [0 Infinity]/D)
Description: The AUC (0-infinity)/D is the area under concentration-time curve extrapolated to infinity postdose normalized by MEDI9929 dose. The PK parameter was estimated based on the serum concentrations of MEDI9929. Serum concentrations of MEDI9929 were measured by enzyme-linked immunosorbent assay.
Time Frame: Predose on Day 1 and Day 2, 4, 7, 11, 15, 22, 29, 43, 57 and 85 post-dose.
Population: PK Population
Measure: Mean (Standard Deviation); unit: μg*day/mL/mg
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Number analyzed (Participants) | 11 | 10
μg*day/mL/mg | 7.27 (2.54) | 6.29 (1.32)

4. Primary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: The PK parameter Cmax was estimated based on the serum concentrations of MEDI9929. Serum concentrations of MEDI9929 were measured by enzyme-linked immunosorbent assay.
Time Frame: Predose on Day 1 and Day 2, 4, 7, 11, 15, 22, 29, 43, 57 and 85 post-dose.
Population: PK Population
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Number analyzed (Participants) | 11 | 10
μg/mL | 24.6 (6.65) | 23.4 (6.82)

5. Primary Outcome: Dose-normalized Cmax (Cmax/D)
Description: The Cmax/D is the maximum observed concentration post dose normalized by MEDI9929 dose. The PK parameter was estimated based on the serum concentrations of MEDI9929. Serum concentrations of MEDI9929 were measured by enzyme-linked immunosorbent assay.
Time Frame: Predose on Day 1 and Day 2, 4, 7, 11, 15, 22, 29, 43, 57 and 85 post-dose.
Population: PK Population
Measure: Mean (Standard Deviation); unit: μg/mL/mg
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Number analyzed (Participants) | 11 | 10
μg/mL/mg | 0.176 (0.0475) | 0.167 (0.0487)

6. Primary Outcome: Time to Reach Cmax (Tmax)
Description: The Tmax is the time to maximum observed serum concentration of MEDI9929. The PK parameter was estimated based on the serum concentrations of MEDI9929. Serum concentrations of MEDI9929 were measured by enzyme-linked immunosorbent assay.
Time Frame: Predose on Day 1 and Day 2, 4, 7, 11, 15, 22, 29, 43, 57 and 85 post-dose.
Population: PK Population
Measure: Median (Full Range); unit: Day
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Number analyzed (Participants) | 11 | 10
Day | 5.98 [0.990 to 9.97] | 4.44 [1.40 to 19.9]

7. Primary Outcome: Terminal Phase Elimination Half Life (t1/2,z)
Description: The t½,z is the time measured for the serum drug concentration of MEDI9929 to decrease by one half. The PK parameter was estimated based on the serum concentrations of MEDI9929. Serum concentrations of MEDI9929 were measured by enzyme-linked immunosorbent assay.
Time Frame: Predose on Day 1 and Day 2, 4, 7, 11, 15, 22, 29, 43, 57 and 85 post-dose.
Population: PK Population
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Number analyzed (Participants) | 11 | 10
Day | 24.0 (4.09) | 26.7 (5.13)

8. Primary Outcome: Apparent Clearance (CL/F)
Description: The PK parameter CL/F was estimated based on the serum concentrations of MEDI9929. Serum concentrations of MEDI9929 were measured by enzyme-linked immunosorbent assay.
Time Frame: Predose on Day 1 and Day 2, 4, 7, 11, 15, 22, 29, 43, 57 and 85 post-dose.
Population: PK Population
Measure: Mean (Standard Deviation); unit: Liter/day
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Number analyzed (Participants) | 11 | 10
Liter/day | 0.153 (0.0507) | 0.166 (0.0376)

9. Primary Outcome: Apparent Steady-state Volume of Distribution (Vss/F)
Description: The PK parameter Vss/F was estimated based on the serum concentrations of MEDI9929. Serum concentrations of MEDI9929 were measured by enzyme-linked immunosorbent assay.
Time Frame: Predose on Day 1 and Day 2, 4, 7, 11, 15, 22, 29, 43, 57 and 85 post-dose.
Population: PK Population
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Number analyzed (Participants) | 11 | 10
Liter | 5.65 (1.60) | 6.55 (2.19)

10. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events
Description: An adverse event (AE) is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious adverse event (SAE) is any AE resulting in any of the following outcomes such as death; initial or prolonged inpatient hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly or birth defect, or is an important medical event that may jeopardize the participant or may require medical intervention to prevent one of the outcomes listed above. A TEAE is defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug. The AEs were summarized using Medical Dictionary for Regulatory Activities version 19.0
Time Frame: From the start of study drug administration up to end of follow-up period, assessed up to Day 85
Population: As-treated Population: All participants who received any treatment of MEDI9929.
Measure: Number; unit: Participants
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Number analyzed (Participants) | 11 | 10
Participants
  Participants with TEAEs | 4 | 4
  Participants with treatment-emergent SAEs | 0 | 0

11. Secondary Outcome: Treatment-emergent Adverse Events Related to Vital Sign Parameters and Physical Findings
Description: Vital signs (blood pressure, temperature, pulse, and respiratory rate) were performed throughout the study. The TEAEs related to vital signs in participants were reported.
Time Frame: From the start of study drug administration up to end of follow-up period, assessed up to Day 85
Population: As-treated Population
Measure: Number; unit: Participants
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Number analyzed (Participants) | 11 | 10
Participants | 0 | 0

12. Secondary Outcome: Treatment-emergent Adverse Events Related to Laboratory Parameters
Description: Laboratory evaluations of blood and urine samples were performed, including hematology (white blood cell count with differential, red blood cell count, hematocrit, hemoglobin and platelet count); serum chemistry: calcium, chloride, potassium, sodium, bicarbonate, aspartate transaminase, alanine transaminase, albumin, uric acid, creatinine, total bilirubin, glucose, alkaline phosphatase, blood urea nitrogen, total protein, and gamma glutamyl transferase; and urinalysis (nitrites, protein, glucose, ketones, urine drug screen, blood, and bilirubin). Number of participants with TEAEs related to laboratory evaluations were reported.
Time Frame: From the start of study drug administration up to end of follow-up period, assessed up to Day 85
Population: As-treated Population
Measure: Number; unit: Participants
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Number analyzed (Participants) | 11 | 10
Participants | 0 | 0

13. Secondary Outcome: Treatment-emergent Adverse Events Related to Electrocardiogram Evaluations
Description: Computerized triplicate 12-lead ECGs as well as Qualitative 12-lead ECGs were obtained during the study. ECG parameters included heart rate, PR, QRS, QT, and corrected QT (QTc) intervals. Number of participants with TEAEs related to ECG after the start of study drug were to be reported.
Time Frame: From the start of study drug administration up to end of follow-up period, assessed up to Day 85
Population: As-treated Population
Measure: Number; unit: Participants
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Number analyzed (Participants) | 11 | 10
Participants | 0 | 0

14. Secondary Outcome: Number of Participants Positive for Anti-drug Antibodies and With Neutralizing Antibodies for MEDI9929 at Any Visit
Description: Blood samples for immunogenicity assessment included the determination of anti-drug antibodies (ADA) for MEDI9929. The incidence rate of positive serum antibodies to MEDI9929 were presented.
Time Frame: Days 1 (predose), 29, 57 and 85
Population: As-treated Population. Neutralizing antibody was tested only for the positive ADA samples. Combined immunogenicity data is presented for all participants (that is 12 to 17 years of age). n= Number of participants analyzed for this outcome measure at the given time point.
Measure: Number; unit: Participants
Groups:
- MEDI9929: On Day 1, a single dose of MEDI9929 was administered subcutaneously to participants, aged 12 to 17 years, inclusive.
Arm/Group | MEDI9929
Number analyzed (Participants) | 21
Participants
  Baseline: ADA positive, n=21 | 1
  Baseline: Positive neutralizing antibody, n=1 | 0
  Post-baseline: ADA positive, n=21 | 1
  Post-baseline: Positive neutralizing antibody, n=1 | 0

ADVERSE EVENTS:
Time Frame: From the start of study drug administration up to end of followup period, assessed up to Day 85.
Arm/Group | MEDI9929, 140 mg, (12 to 14 Years) | MEDI9929, 140 mg, (15 to 17 Years)
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 4/11 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI9929, 140 mg, (12 to 14 Years) (N=11) | MEDI9929, 140 mg, (15 to 17 Years) (N=10)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.